CLINICAL TRIAL: NCT06800430
Title: Vein Graft Failure and Cardiovascular Consequences of Coronary Artery Bypass Graft Surgery
Brief Title: Graft Failure and Consequences of Coronary Artery Bypass Graft Surgery
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC24158; SS/CH/09/002 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2025-01-22; First posted 2025-01-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Bypass; Graft Failure; Coronary Artery Bypass Graft; Coronary Artery Bypass Graft Surgery (CABG)
Keywords: CABG; graft failure; coronary artery bypass; cardiovascular; heart surgery; cardiac surgery; coronary artery bypass graft; cardiovascular disease; heart disease; positron emission tomography
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Ga(III)-DOTATOC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples (up to 60ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Patients undergoing CABG surgery: 40 patients (maximum 120) undergoing CABG surgery with multi-vessel disease and at least one saphenous vein graft.
  Interventions: Radiation: Hybrid [18F]-GP1, [68Ga]-DOTATATE, [68Ga]-FAPI total-body positron emission tomography and coronary computed tomography coronary angiography
- Cohort 2: Patients with symptomatic saphenous vein graft vasculopathy: 30 patients with prior CABG surgery (at least 5 years previously) with multi-vessel disease and two or more saphenous vein grafts, who have been referred for invasive coronary angiography due to symptoms and with a high suspicion of graft vasculopathy.
  Interventions: Radiation: Hybrid [18F]-GP1, [68Ga]-DOTATATE, [68Ga]-FAPI total-body positron emission tomography and coronary computed tomography coronary angiography

INTERVENTIONS:
Radiation: Hybrid [18F]-GP1, [68Ga]-DOTATATE, [68Ga]-FAPI total-body positron emission tomography and coronary computed tomography coronary angiography — Patients undergo hybrid [18F]-GP1, [68Ga]-FAPI and [68Ga]-DOTATATE total body PET-CT imaging (Biograph Vision Quadra, Siemens) and contrast-enhanced electrocardiogram gated CT coronary angiogram (CTCA), within 28 days (+/- 28 days) of their CABG surgery and again at 12 month follow-up.
  Groups: Cohort 1: Patients undergoing CABG surgery
Radiation: Hybrid [18F]-GP1, [68Ga]-DOTATATE, [68Ga]-FAPI total-body positron emission tomography and coronary computed tomography coronary angiography — Patients undergo hybrid [18F]-GP1, [68Ga]-FAPI and [68Ga]-DOTATATE total body PET-CT imaging (Biograph Vision Quadra, Siemens) and contrast-enhanced electrocardiogram gated CT coronary angiogram (CTCA), prior to their clinical invasive coronary angiography.
  Groups: Cohort 2: Patients with symptomatic saphenous vein graft vasculopathy

SUMMARY:
Coronary artery bypass graft (CABG) surgery is the commonest type of heart operation performed. During this, arteries or veins (termed 'grafts') are used to supply blood around blockages within the blood vessels that supply the heart. Unfortunately, these grafts can sometimes fail, and patients can also experience complications like heart attacks and strokes, after surgery. It is known that vein grafts are more likely to narrow over time. Additionally, treating vein graft failure is very challenging, as repeat surgery is riskier and procedures to stent open the veins can also fail. However, it is not fully understood why these complications occur.

In this study, the investigators will use an imaging technique called a total-body Positron Emission Tomography (PET) scan. This uses special radioactive dyes (radiotracers) to look at what is happening inside vein grafts. With this technique, the investigators will also be able to see what is happening to the heart, brain and wider parts of the body after CABG surgery.

This study will aim to recruit 70 participants in total (maximum 150). 40 (maximum of 120) of these participants will have recently undergone CABG surgery and received ≥1 vein graft. The remaining 30 will have undergone CABG surgery ≥5 years ago and will have symptoms suggestive of vein graft failure.

The study will last a total of 36 months and will involve participants undertaking the following assessments:

1. Total-body Positron Emission Tomography and Computed Tomography (PET-CT) scan
2. Ultrasound scan of the heart (echocardiogram)
3. A blood test - up to four tablespoons (60 mL) of blood will be taken for immediate testing and the remainder will be stored for future ethically approved studies.

DETAILED DESCRIPTION:
This is an observational cohort study investigating the role of inflammation, thrombosis and fibrosis in saphenous vein graft failure following CABG surgery. The presence and distribution of these processes will be examined in one cohort overtime (immediately following surgery and at 1 year-follow up) and at one time-point in a second cohort with clinically suspected vein graft failure.

Participants in both cohorts will undergo clinical review (including blood sampling), transthoracic echocardiogram and combined total-body positron emission tomography computed tomography (PET-CT) imaging, with CT coronary angiography.

ELIGIBILITY:
INCLUSION CRITERIA:

Cohort 1: Patients undergoing CABG surgery

* Males and females over 18 years of age
* Patients undergoing CABG surgery for multivessel coronary artery disease, who receive at least one saphenous vein graft

Cohort 2: Patients with symptomatic saphenous vein graft vasculopathy

* Males and females over 18 years of age
* Patients who underwent CABG surgery ≥ 5 years prior to recruitment for multivessel disease and received 2 or more saphenous vein grafts
* Referred for invasive coronary angiography due to recurrent symptoms and with a high suspicion of graft vasculopathy

EXCLUSION CRITERIA:

* Patients with a life expectancy of < 2 years
* Renal failure (estimated glomerular filtration rate <30 mL/min/1.73 m2)
* Patients on immunosuppressive therapies
* Females of child-bearing age who are pregnant or breastfeeding,
* Known allergy or contraindications to iodinated contrast or radiotracer
* Patients who are unable to tolerate the supine position
* Patients who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit two populations of patients following CABG surgery. Participants will be prospectively recruited following CABG surgery (cohort 1), or identification of clinically suspected saphenous vein graft failure (cohort 2). Recruitment will for both cohorts will be from a single, tertiary centre (Royal Infirmary of Edinburgh).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-08-06 (Estimated)

PRIMARY OUTCOMES:
Platelet activation | 3 years
  The degree and location of platelet activation within saphenous vein grafts, measured using standard uptake values and tissue-to-background ratios of [18F]-GP1.
Fibroblast activation | 3 years
  The degree and location of fibroblast activation within saphenous vein grafts, measured using standard uptake values and tissue-to-background ratios of [68Ga]-FAPI.
Macrophage activation | 3 years
  The degree and location of macrophage activation within saphenous vein grafts, measured using standard uptake values and tissue-to-background ratios of [68Ga]-DOTATATE.

SECONDARY OUTCOMES:
Systemic cardiovascular disease | 3 years
  The secondary endpoints will include the presence of systemic thrombotic, fibrotic or inflammatory cardiovascular disease, assessed through biomarker and CT imaging analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No